CLINICAL TRIAL: NCT01256697
Title: The Effect of Oral Administration of 9-cis Rich Powder of the Alga Dunaliella
Brief Title: The Effect of Oral Administration of 9-cis Rich Powder of the Alga Dunaliella Bardawil on Visual Functions im Patients With Retinitis Pigmentosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ygal Rotenstreich, Ophthalmologist, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA -08-5086-YR-CTIL
Record Dates: First submitted 2010-02-25; First posted 2010-12-08 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alga Dunaliella Bardawil (Experimental)
  Interventions: Dietary Supplement: Alga Dunaliella Bardawil; Dietary Supplement: Alga Dunaliella Bardawill
- Sugar pill (Placebo Comparator)
  Interventions: Other: Sugar pill

INTERVENTIONS:
Dietary Supplement: Alga Dunaliella Bardawil — 9-cis Rich Powder
  Arms: Alga Dunaliella Bardawil
Dietary Supplement: Alga Dunaliella Bardawill — 9-cis Rich Powder
  Arms: Alga Dunaliella Bardawil
Other: Sugar pill — Sugar pill
  Arms: Sugar pill

SUMMARY:
Retinitis pigmentosa is a genetically determined disease consisting of progressive centripetal retinal degeneration starting in the rods outer segments. Its prevalence is 1:4000 people and is the fourth most common blinding disease in Israel in 2004 [7% of all blindness]. The investigators tried to treat a non-progressive form of the disease [Fundus Albipunctatus] by oral therapy of the food supplement made from alga Dunaliella bardawil composed of approximately 50% 9-cis β-carotene. The alga Dunaliella bardawil accumulates high concentration of β -carotene when grown under appropriate conditions. The β -carotene of the alga is composed of approximately 50% of all-trans - β carotene and 50% 9-cis β -carotene.

The 9-cis β -carotene has shown to be a precursor of 9-cis retinoic acid both in-vitro in human intestinal mucosa and in-vivo in a ferret, perfuse with 9-cis b-carotene. The night vision, as measured objectively by electroretinography (ERG) more than doubled in six patients tested. The visual field was also improved significantly.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study.
* Men or women aged 18 years or older.
* Electroretinogram (ERG) responses compatible with the diagnosis of Retinitis Pigmentosa

Exclusion Criteria:

* Current smokers.
* Current use of Vitamin A/ beta carotene supplements.
* Active arterial disease within 3 months of study entry such as unstable angina, myocardial infarction, transient ischemic attack (TIA), stroke, and coronary artery bypass graft (CABG) surgery.
* History of malignancy, except basal or squamous cell skin carcinoma.
* Pregnant women, women who are breast feeding, and women of childbearing potential who are not using chemical or mechanical contraception.
* Uncontrolled hypertension defined as either resting diastolic blood pressure of >95mmHg (taken from the mean of 3 readings) or resting systolic blood Pressure of > 180 mmHg.
* History of alcohol abuse or drug abuse, or both.
* Patient plans to engage in vigorous exercise or an aggressive diet regimen.
* Uncontrolled endocrine or metabolic disease.
* Participation in another investigational drug study within 4 weeks of entry into this study.
* Serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
* Subject whose hormone replacement therapy (HRT) or oral contraceptive therapy (OCT) was initiated within the 3 month prior to enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Electroretinogram scotopic maxiamal b-wave amplitude responses in microvolts | 1 year
  Using the protocol of the International Society for Clinical Electrophysiology of Vision and the UTAS 3000 system (LKC Technologies, Gaithersburg, MD), we recorded full-field electroretinographic responses from both eyes of each patient. The scotopic conditions, after 30 minutes of dark adaptation we recorded the maximal scotopic response. The b-wave amplitude responses will be messured in each eye.

SECONDARY OUTCOMES:
The area within the Dark adapted chromatic Goldamann Visual field in isopters in cm2 | 1 year
  Kinetic visual field for chromatic stimuli will be recorded in both eye after 30 minutes of dark adaptation. area of vision within the isopter will be measured by software in cm2.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Result] Rotenstreich Y, Belkin M, Sadetzki S, Chetrit A, Ferman-Attar G, Sher I, Harari A, Shaish A, Harats D. Treatment with 9-cis beta-carotene-rich powder in patients with retinitis pigmentosa: a randomized crossover trial. JAMA Ophthalmol. 2013 Aug;131(8):985-92. doi: 10.1001/jamaophthalmol.2013.147. PMID 23700011
- [Derived] Schwartz SG, Wang X, Chavis P, Kuriyan AE, Abariga SA. Vitamin A and fish oils for preventing the progression of retinitis pigmentosa. Cochrane Database Syst Rev. 2020 Jun 18;6(6):CD008428. doi: 10.1002/14651858.CD008428.pub3. PMID 32573764